CLINICAL TRIAL: NCT05655806
Title: Effect of Aminophylline Bolus Versus Infusion on Recovery Time in Patients Undergoing Lumbar Spine Surgery: Double Blind Randomized Controlled Trial
Brief Title: Effect of Aminophylline Bolus Versus Infusion on Recovery Time in Patients Undergoing Lumbar Spine Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hussein Sayed Hasan, lecturer of anesthesia , surgical ICU and pain managment, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-56-2022/MD
Record Dates: First submitted 2022-11-14; First posted 2022-12-19 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Anesthesia
Keywords: aminophylline; recovery time; time of extubation
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: drugs will be prepared by another person who is not giving drugs or collecting data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): will receive aminophylline loading dose 5mg/kg on a 50 cm syringe using syringe pump over 5 minutes and maintenance dose 1.5 mg/kg/hr as a continuous infusion half an hour before discontinuation of isoflurane, and after discontinuation of isoflurane a 5 cm syringe of saline will be given over 5 minutes
  Interventions: Drug: Aminophylline bolus then infusion
- group B (Active Comparator): will receive a 50 cm syringe of saline using syringe pump over 5 minutes and maintenance continuous infusion of saline half an hour before discontinuation of isoflurane, and after discontinuation of isoflurane a 5cm syringe of aminophylline bolus 5mg\kg will be given over 5 minutes
  Interventions: Drug: aminophylline bolus
- group C (Placebo Comparator): will receive a 50 cm syringe of saline using syringe pump over 5 minutes and maintenance continuous infusion of saline half an hour before discontinuation of isoflurane, and after discontinuation of isoflurane a 5 cm syringe of saline will be given
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Aminophylline bolus then infusion — half an hour before discontinuation of isoflurane
  Arms: group A
Drug: aminophylline bolus — after discontinuation of isoflurane
  Arms: group B
Drug: normal saline — given as placebo
  Arms: group C

SUMMARY:
To determine optimal dose, method and time of administration of aminophylline to enhance the recovery from general anesthesia.

andTo estimate the recovery time from isoflurane closure in each group. We hypothesize that starting administration of loading and maintenance dose of aminophylline half an hour before discontinuing isoflurane will shorten the duration needed to extubate patients undergoing lumbar disc surgery. We hypothesized that it will yield superior results compared to bolus administration after discontinuing isoflurane.

DETAILED DESCRIPTION:
* it is a randomized double blinded study
* Population of study:

Adult male and female patients undergoing single or double level lumbar disc laminectomy, discectomy and /or fixation.

recruitment of cases will be started after getting approval of ethical committee in our faculty (done and its number is N-56-2022/MD) and registration in clinicaltrials.gov and getting a unique number

- Study location: This study will be set at neurosurgery theater, kasr alainy Hospital, Cairo University.

* Methodology in details: On arrival to the operating room, standard monitoring equipment will be applied, including electrocardiography (ECG), automated non-invasive blood pressure (NIBP), pulse oximetry and baseline readings will be recorded. Peripheral IV access will be inserted. Antibiotic and antiemetic will be given preoperatively. Entropy (GE Entropy healthcare) monitoring which is a valuable tool for measuring depth of anesthesia will be used, Response entropy (RE) and state entropy (SE) will be monitored using specific entropy sensors that will be placed on the patient's forehead according to the manufacturer's instructions.
* No sedative premedication will be given. Induction of general anesthesia will be done by propofol 2-3mg/kg, fentanyl 2ug/kg and endotracheal intubation will be facilitated by atracurium 0.5 mg/kg. Anesthesia will be maintained by isoflurane 1.2 % and atracurium 0.1 mg/kg/30min, morphine 0.1 mg/kg I.V will be given for intra and post -operative analgesia .Near the end of the end of the surgery, the study population will be randomized to three groups.
* . Group A will receive aminophylline loading dose 5mg/kg on a 50 cm syringe using syringe pump over 5 minutes and maintenance dose 1.5 mg/kg/hr as a continuous infusion half an hour before discontinuation of isoflurane, and after discontinuation of isoflurane a 5 cm syringe of saline will be given over 5 minutes . Group B will receive a 50 cm syringe of saline using syringe pump over 5 minutes and maintenance continuous infusion of saline half an hour before discontinuation of isoflurane, and after discontinuation of isoflurane a 5cm syringe of aminophylline bolus 5mg\kg will be given over 5 minutes. On the other hand, group C will receive a 50 cm syringe of saline using syringe pump over 5 minutes and maintenance continuous infusion of saline half an hour before discontinuation of isoflurane, and after discontinuation of isoflurane a 5 cm syringe of saline will be given. These syringes will be prepared by an independent anesthesiologist and contain either aminophylline or a similar volume of normal saline. Recovery and data collection will be assessed by a second anesthesiologist who will not be aware of the group to which the patient will be allocated, also the patients will not know to which group they will be allocated. Entropy values, heart rate, blood pressure will be monitored in all patients before and every 5 minutes after injection of the test drug till half an hour after extubation. The following variables will be measured in all groups eye -opening in response to vocal request and time to extubation after discontinuation of anesthetic agent.
* Entropy will be used to monitor the depth of anesthesia using frontal electromyography through measuring irregularity of signals. High entropy values indicate high irregularity of signals which signifies that the patient is awake. A more regular signal produce low entropy values which can be associated with low probability of consciousness, so we will use it to assess the speed of return of conscious level after discontinuation of isoflurane.
* At the end of surgery, anesthetic gases will be discontinued and patients will be ventilated with 100% O2. For the antagonism of muscle relaxation, neostigmine 0.05mg/kg and atropine 0.01mg/kg will be given

sample size :

Power analysis was performed using one-way ANOVA test to detect at least 20% difference in time to extubation as the primary outcome of our study. Based on previous study(10); the mean ± SD time to extubation in the single shot aminophylline group was 6.6 ± 2.47 minutes.

At an α error of 0.05 and power of 0.8. A minimum of 93 patients was calculated. The sample will be increased 99 patients (33 patients per arm) for the possible dropouts. Sample size was calculated using G*Power 3 software.

11- Statistical analysis

The statistical package for the social sciences version 23 (SPSS, Inc, Chicago, IL, USA) will be used for statistical analysis. Descriptive statistics will be done for quantitative data by mean & standard deviation (SD), while they are done for categorical data by number and percentage. Studies will be done to calculate the inter and intra-observer variability. The level of significance is taken at P value<0.05 to exclude false positive results

ELIGIBILITY:
Inclusion Criteria:

ASA I-II. 20-50 years old patients. Both sexes Patients undergoing single or double level lumbar laminectomy ,discectomy and/or fixation

Exclusion Criteria:

Contraindications to the use of aminophylline as cardiac patients, patients with renal impairment, hepatic dysfunction, hypo or hyperthyroidism and epilepsy.

Patients who have hypersensitivity to aminophylline Emergency operations. Operative time exceeding 5 hours

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Recovery time | one hour
  Time to extubation from closure of isoflurane to extubation in minutes

SECONDARY OUTCOMES:
Response entropy (RE) | 4 hours
  after induction of anesthesia, every 30 minutes throughout the operation and every 5 minutes after injection of the test drug and till half an hour after extubation
State entropy (SE) | 4 hours
  after induction of anesthesia, every 30 minutes throughout the operation, every 5minutes after injection of the test drug half an hour after extubation.
Mean arterial blood pressure | 4 hours
  base line after induction of anesthesia, every 30 minutes throughout the operation, every 5 minutes after injection of the test drug and half an hour after extubation.
heart rate | 4 hours
  base line after induction of anesthesia, every 30 minutes throughout the operation, every 5 minutes after injection of the test drug and half an hour after extubation.
The total dose of aminophylline | two hours
  in mg in groups A and B
The incidence of side effects | 24 hours
  as chest pain ,fainting, persistent vomiting, rapid pulse, arrhythmias and seizure within 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El Tahan MR. Effects of aminophylline on cognitive recovery after sevoflurane anesthesia. J Anesth. 2011 Oct;25(5):648-56. doi: 10.1007/s00540-011-1190-8. Epub 2011 Jul 14. PMID 21755342
- [Background] Elsarrag M, Soldozy S, Patel P, Norat P, Sokolowski JD, Park MS, Tvrdik P, Kalani MYS. Enhanced recovery after spine surgery: a systematic review. Neurosurg Focus. 2019 Apr 1;46(4):E3. doi: 10.3171/2019.1.FOCUS18700. PMID 30933920
- [Background] Wang Q, Fong R, Mason P, Fox AP, Xie Z. Caffeine accelerates recovery from general anesthesia. J Neurophysiol. 2014 Mar;111(6):1331-40. doi: 10.1152/jn.00792.2013. Epub 2013 Dec 26. PMID 24375022
- [Background] Ghaffaripour S, Khosravi MB, Rahimi A, Sahmedini MA, Chohedri A, Mahmoudi H, Kazemi MR. The effects of Aminophylline on clinical recovery and bispectral index in patients anesthetized with total intravenous anaesthesia. Pak J Med Sci. 2014 Nov-Dec;30(6):1351-5. doi: 10.12669/pjms.306.5853. PMID 25674137
- [Background] Wang HL, Tang SH, Wang XQ, Gong WH, Liu XM, Lei WF. Doxapram hastens the recovery following total intravenous anesthesia with dexmedetomidine, propofol and remifentanil. Exp Ther Med. 2015 Apr;9(4):1518-1522. doi: 10.3892/etm.2015.2249. Epub 2015 Feb 2. PMID 25780462